CLINICAL TRIAL: NCT05226858
Title: Emergency Physician Performed Transesophageal Echocardiography To Diagnose Blunt Traumatic Aortic Injury
Brief Title: Transesophageal Echocardiography To Diagnose Blunt Traumatic Aortic Injury Traumatic Aortic Injury
Status: Recruiting | Type: Observational
Sponsor: Hospital Raja Permaisuri Bainun (Other Government)
Collaborators: Hospital Sultanah Bahiyah (Other Government); Kuala Lumpur General Hospital (Other Government); Hospital Melaka (Unknown); Hospital Queen Elizabeth, Malaysia (Other Government); University of Malaya (Other)
Responsible Party: Principal Investigator, Dr. Adi Bin Osman, Principal Investigator, Hospital Raja Permaisuri Bainun
Other Study IDs: NMRR-21-518-59250 (IIR)
Record Dates: First submitted 2022-01-04; First posted 2022-02-07 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Trauma Chest
Keywords: Transesophageal echocardiography; Aorta; Trauma; Emergency department; Blunt Trauma
MeSH Terms: conditions — Thoracic Injuries; Wounds and Injuries; Emergencies; Wounds, Nonpenetrating | interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trauma patients with suspected blunt traumatic aortic injury (BTAI): All trauma patients with suspected BTAI at the emergency department who require both transesophageal echocardiography (TEE) and computed tomography angiography (CTA).
  Interventions: Diagnostic Test: Transesophageal echocardiography (TEE)

INTERVENTIONS:
Diagnostic Test: Transesophageal echocardiography (TEE) — Sensitivity and specificity of TEE in identification of BTAI

SUMMARY:
To determine test performance of transesophageal echocardiography performed by emergency physician ultrasound for the identification of blunt traumatic aortic injury in chest trauma.

DETAILED DESCRIPTION:
This is a multicentre prospective observational trial. All trauma patients with suspected BTAI at the emergency department (ED) will undergo resuscitative transesophageal echocardiography to evaluate the thoracic aorta.

Resuscitative TEE is a minimally invasive procedure to evaluate all chest trauma patients. Besides the aorta, TEE can also provide other useful information regarding the hemodynamic status, cardiac function and lung pathology of the patient.

Patients will be recruited into the study by investigators who take informed consent from the patient or next of kin prior to the TEE procedure.

For all patients with suspected BTAI, CTA is mandatory to confirm the diagnosis of BTAI.

TEE findings of BTAI will be compared to CTA which will be considered the reference standard unless confirmation is available from surgical procedures or autopsy.

Inter-observer variability for normal or pathological TEE images interpretation is performed prior to the initiation of the study.

ELIGIBILITY:
Inclusion Criteria:

All trauma patients with suspected BTAI in the emergency department (ED) who undergo both TEE and CTA.

Exclusion Criteria:

1. Children (age under 18 years) will not be eligible for inclusion in this study.
2. Patients with contraindication to TEE such as suspected esophageal injury or pathology

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suspected BTAI are defined by the presence of at least one of the following criteria
  1. high risk mechanism of injury (deceleration or crush injury),
  2. clinical findings (external chest trauma or unexplained hypotension) or
  3. chest Xray findings suspicious of BTAI (mediastinal widening, a blurred aortic knob, apical capping of the lung, a depressed left bronchus, a displaced nasogastric, mediastinal widening, or fractured first or second ribs).
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of TEE in identification of BTAI | 1 year
  To determine the test performance of transesophageal echocardiography in the identification of BTAI in comparison to CTA.

CONTACTS AND LOCATIONS:
Overall Officials: Adi Osman, MD, Principal Investigator — Hospital Raja Permaisuri Bainun
Locations (6):
- Malaysia (6):
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Hospital Queen Elizabeth, Kota Kinabalu, Sabah
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University of Malaya, Kuala Lumpur
  - Hospital Melaka, Malacca

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/58/NCT05226858/Prot_SAP_001.pdf